CLINICAL TRIAL: NCT01241617
Title: Randomized Trial Between Buttressed and Non Buttressed Stapling in Pulmonary Lobectomy
Brief Title: ENDO GIA Stapler With Duet Tissue Reinforcement System (TRS) Used in Pulmonary Resections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covidien is conducting a voluntary recall of DuetTRS™ use in the thoracic cavity. IFU is revised to contraindicate use in adult and pediatric thoracic surgeries
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Juntendo-530
Record Dates: First submitted 2010-07-30; First posted 2010-11-16 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Lung Disease
Keywords: Lung disease; Lobectomy; Pulmonary resection
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duet TRS (Active Comparator): Endo GIA with integrated Duet TRS
  Interventions: Device: Duet TRS
- Endo GIA (Active Comparator): Endo GIA stapler with Single Use Loading units
  Interventions: Device: Endo GIA

INTERVENTIONS:
Device: Duet TRS — Endo GIA stapler with integrated Duet TRS
  Other Names: Endo GIA stapler with integrated Duet TRS
  Arms: Duet TRS
Device: Endo GIA — Endo GIA stapler with Single Use Loading Units
  Other Names: Endo GIA stapler with Single Use Loading Units
  Arms: Endo GIA

SUMMARY:
The objective of this study is to confirm superiority between a test treatment group using Endo GIA stapler with Duet Tissue Reinforcement System (TRS) and a current international standard of care group using a conventional stapler in patients undergoing pulmonary lobectomy surgery, using a randomized comparative study of the frequency of intraoperative air leak.

DETAILED DESCRIPTION:
Air leak is a complication of pulmonary surgical procedures that include pulmonary lobectomy, segmentectomy, and bullectomy, reported to occur in 33% to 75% of cases.

Prolonged air leak continuing for more than 7 days is reported to have a prevalence of greater than 15%. The presence of a history of smoking, preoperative steroid use, emphysema, low pulmonary function, pleural adhesion, and apical lung wedge resection are shown to be risk factors for prolonged air leak which lengthens the duration of drain placement, increases the days of hospitalization, and reduces patient ADL and QOL. Prolonged air leak may also result in serious complications, such as empyema.

Tissue reinforcement materials widely used as a pleural reinforcement to prevent air leaks during lung surgery, and are reported as a safe and effective material for body tissue reinforcement. Covidien Japan Inc. has developed a surgical stapler (Endo GIA Duet TRS) with an attached reinforcement material. This study will investigate the reinforcement effect on the staple line of using the newly developed surgical stapler with an attached reinforcement material.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 20-79 years of age.
* The patient is eligible to be given pulmonary Lobectomy.
* The patient is scheduled to undergo pulmonary Lobectomy.
* Performance status 0~1 (Eastern Cooperative Oncology Group classification).
* The patient has no history of lung surgery.
* The patient is healthy organ function.
* The patient is scheduled for surgery with staplers .
* The patient must be willing and able to participate in the study procedures and able to understand and sign the informed consent.

Exclusion Criteria:

* The patient has suffered thoracic trauma or has previously undergone pneumonectomy surgery.
* The patient has an active bacterial infection or fungal infection.
* The patient is undergoing continuing systemic administration (intravenous or oral) of steroids.
* The patient condition is complicated by uncontrolled diabetes mellitus.
* The patient participation is judged difficult due to study complications related to a psychiatric disorder or psychological symptoms.
* The patient undergoes surgical procedure other than lobectomy during surgery.
* Reinforcement material other than the study materials are applied during surgery.
* The patient judged unsuitable for study participation by the investigator for any other reason.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Frequency of intraoperative air leak | Day 0
  Occurence of intraoperative air leak will vary from patient to patient and will be recorded for all patients.

SECONDARY OUTCOMES:
Postoperative duration of air leak | Month 1 (Average time period)
  Duration of air leak will vary from patient to patient. Published literature states a duration of greater than 7 days occurs in 15% of patients.
Duration of chest drainage | Month 1 (Average time period)
  Duration of chest drainage will vary from patient to patient.
Frequency of intraoperative sealant use | Day 0
  The need to use a sealant intraoperatively will be assessed for each patient during surgery.
Incidence of intraoperative adverse events | Day 0
  The occurence of adverse events during surgery will be recorded for each patient.
Incidence of postoperative adverse events | Month 1 (Average time period)
  Patients are not required to return to the clinic at a specific time point. Any adverse events that occur after discharge will be captured.
Days of hospitalization | Month 1 (Average time period)
  Discharge date will vary from patient to patient

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Suzuki, MD, Principal Investigator — Juntendo University
Locations (1):
- Junendo University School of Medicine, Tokyo, Japan